CLINICAL TRIAL: NCT00273559
Title: A Single Center, Open Label, Comparative, Controlled Trial to Assess the Risks and Benefits of Steroid Elimination vs. Steroid Therapy After Renal Transplantation
Brief Title: A Study Comparing Outcomes of Kidney Transplants in Patients on Steroids Versus Those Who Discontinue Steroids
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Florida Hospital Transplant Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Novartis (Industry)
Responsible Party: Michael Angelis, MD, Florida Hospital Transplant Center
Other Study IDs: TL092005-1
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2007-11

CONDITIONS: Kidney Diseases
Keywords: Renal Transplantation
MeSH Terms: conditions — Kidney Diseases | interventions — Prednisone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: subjects who remain on steroids after discharge
- 2: Subjects will be off steroids at the time of discharge
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: prednisone — group 2 will remain on 5 mg of prednisone for at least 90 days post transplant.
  Groups: 2

SUMMARY:
The purpose of this study is to compare the risks and benefits of steroid elimination versus steroid therapy in renal transplant patients particularly looking at the effects on bone mass, lipids, hypertension, and new onset diabetes.

DETAILED DESCRIPTION:
The use of steroids after renal transplantation has been invaluable, resulting in higher rates of long term survival of the transplanted kidney. However, post-operative steroids are also associated with frequent post-operative and long term complications. There have been steroid elimination studies analyzing acute rejection rates, graft and patient survival. These studies show that many patients can safely have steroids withdrawn with equivalent results whan compared to those who remain on steroids.

With this study we will be using a rapid steroid elimination protocol for 40 patients and compare 20 patients who remain on steroids. We hope to show a decreased rate of complications such as osteopenia/osteoporosis, new onset diabetes, and a decrease in cardiovascular risk factors such as hyperlipidemia and hypertension.

Solumedrol will be given to all patients at the time of transplant followed by a prednisone taper. Those remaining on steroids will be discharged on prednisone 5 mg daily. Those in whom steroids are eliminated will be off prednisone by discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a single renal transplant from deceased or living donor
* Adults 18 years and older
* First or second renal transplant
* Capable of understanding the purposes of the study, has given written informed consent, and agrees to comply with the study requirements
* Women of child bearing age should have a negative serum pregnancy test

Exclusion Criteria:

* Greater than 2 renal transplants
* Age < 18 years
* Patients receiving immunosuppressive therapy within the preceding 28 days for first transplant and 3 months for the second transplant
* Cold ischemia time > 30 hours
* History of malignancy in the last 5 years except successfully treated localized non-melanoma skin cancer
* HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV) positive serology
* Loss of previous transplant in < 1 year
* History of non-compliance
* Any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may impair communication with the investigator or compliance with study procedures
* Multiple organ transplant
* History of chronic steroid use except for inhaled steroids for asthma
* Pregnant or lactating females
* Women of childbearing potential not willing to use a reliable form of contraception.
* Patients with severe medical condition(s) that, in the view of the investigator, prohibits participation in the study
* Known sensitivity to study drugs or class of study drugs
* Use of any investigational agent in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: de novo renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Acute rejection | 6 months
Patient and graft survival | 6 months
Incidence of infection | one year

SECONDARY OUTCOMES:
Quality of life (health survey) | one year
Incidence of post-transplant diabetes | one year
Incidence of osteopenia/osteoporosis at baseline and one year | one year
Renal function | one year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Angelis, MD, Principal Investigator — Florida Hospital Transplant Center
Locations (1):
- Florida Hospital Transplant Center, Orlando, Florida, United States